CLINICAL TRIAL: NCT03344276
Title: Assessing Neurocognition After Cerebrovascular Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Alexander A. Khalessi MD MS FAANS, Acting Clinical Chief UCSD, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170103
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Carotid Artery Diseases; Neurocognitive Dysfunction
Keywords: carotid stenosis; neurocognition; carotid stenting; circle of willis
MeSH Terms: conditions — Carotid Artery Diseases; Cognition Disorders; Carotid Stenosis

STUDY DESIGN:
Intervention Model Description: In this pilot study 20 patients, undergoing CAS for CS, will undergo cognitive testing at 2 time points before intervention (1 months, and 2 months) and at 2 time points after invention (1 month and 2 months). The two preoperative time points will serve as the control group and the two postoperative time points will serve as the intervention group.
  Patients will serve as their own controls, classifying the study as a within-subjects design. Patients will also have venous blood drawn to ascertain the change in serum markers associated with endothelial dysfunction and inflammation before and after intervention. Finally, patients will have magnetic resonance imaging (MRA) one month before intervention and 2 months after intervention in order to assess changes in global cerebral blood flow.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (Active Comparator): Patients, as outlined by NASCET criteria, will have between 50 symptomatic stenosis or 70% asymptomatic stenosis of the carotid artery. Patients, undergoing carotid artery stenting for carotid stenosis, will undergo cognitive testing at 2 time points before intervention (1 months, and 2 months). The two preoperative time points will serve as the control group.
  Interventions: Diagnostic Test: Neurocognitive Assessments; Diagnostic Test: Measurements of inflammatory biomarkers
- Intervention Group (Experimental): Patients, as outlined by NASCET criteria, will have between 50 symptomatic stenosis or 70% asymptomatic stenosis of the carotid artery. Patients, undergoing carotid artery stenting for carotid stenosis, will undergo cognitive testing at 2 time points after invention (1 month and 2 months). The two postoperative time points will serve as the intervention group.
  Interventions: Diagnostic Test: Neurocognitive Assessments; Diagnostic Test: Measurements of inflammatory biomarkers; Procedure: Carotid Artery Stenting

INTERVENTIONS:
Diagnostic Test: Neurocognitive Assessments — Patients will undergo carotid artery stenting for 50-70% carotid artery stenosis. Prior to surgery patients will undergo a battery of neurocogntive assessments 1 month and 2 months prior to surgery.
Diagnostic Test: Measurements of inflammatory biomarkers — Patients will undergo carotid artery stenting for 50-70% carotid artery stenosis. After surgery, patients will undergo blood draws to measure for inflammatory biomarkers.
Procedure: Carotid Artery Stenting — Patients will undergo carotid artery stenting for 50-70% carotid artery stenosis.
  Arms: Intervention Group

SUMMARY:
Decreased blood flow to the brain can cause decreased cognitive function. Carotid disease can result in decreased blood flow to the brain. The investigators seek to assess this relationship prospectively through performing a battery of neurocognitive assessments, collection of serum markers of inflammation, and through neuroimaging at two points before intervention (2 months and 1 month before stenting) and at two points after intervention (1 month and 2 months after intervention). The goal is to provide prospective evidence to identify the extent to which carotid stenosis and hypoperfusion of the brain results in diminished neurocognitive performance, and see if serum biomarkers before and after stenting correlate with these findings.

DETAILED DESCRIPTION:
Patients are being asked to partake in this study because the PI has decided on clinical grounds as outlined in the clinical trial, NASCET, (either asymptomatic 70% carotid stenosis or symptomatic >50% carotid stenosis) that CAS or CEA is indicated. The only aspect of the study that is research is the cognitive testing, the inflammatory blood markers, and components of the neuroimaging.

In this pilot study 20 patients, undergoing CAS for CS, will undergo cognitive testing at 2 time points before intervention (1 months, and 2 months) and at 2 time points after invention (1 month and 2 months). The two preoperative time points will serve as the control group and the two postoperative time points will serve as the intervention group.

Patients, as outlined by NASCET criteria, will have between 50% symptomatic stenosis or 70% asymptomatic stenosis of the carotid artery. If patients present acutely or are otherwise clinically determined to be unstable (e.g. crescendo TIAs, intolerance of normal physiologic blood pressure, etc.) due to their carotid disease, they will excluded from the study.

Patients will serve as their own controls, classifying the study as a within-subjects design. Patients will also have venous blood drawn to ascertain the change in serum markers associated with endothelial dysfunction and inflammation before and after intervention. Finally, patients will have magnetic resonance imaging (MRA) one month before intervention and 2 months after intervention in order to assess changes in global cerebral blood flow.

The following neurocognitive tests will take place - the duration of all typically takes one hour to complete.

1. Memory measured with the Hopkins Verbal Learning Test-Revised (HVLT-R) and Rey Complex Figure
2. Executive function assessed with Trails A and B
3. Attention/processing speed measured with Wechsler Adult Intelligence Scale Digit Span and Coding subtests
4. Language assessed with the Multilingual Naming Test and Verbal Fluency
5. Visuospatial abilities measured with Block Design
6. Global cognition measured with Mattis Dementia Rating Scale
7. Estimated premorbid intelligence measured with the American version of the National Adult Reading Test (preoperatively only)
8. Mood assessed with the Beck Depression Inventory-II (BDI-II) and Beck Anxiety Inventory (BAI) Biomarkers, as a proxy for systemic inflammation will also be collected. The following biomarkers are associated with inflammation-TNF-α, IL-6, IL-1β, CRP, IFN-γ and endothelial cell activation-sICAM sVCAM will be obtained from venous blood (5 ml) and stored at -80° C until the time of electrochemiluminescence assay. As an accompanying measurement of inflammation, complete blood counts will be assessed.

R statistical software will be used for the statistical analysis. Fisher exact, chi square, and logistic regression testing will be used to assess categorical data while paired t tests and linear regression models will be used to assess continuous variables. Multivariable univariate logistic and linear regression will be performed to assess if carotid intervention is associated with statistically significant changes in neurocognitive performance or changes in serum biomarker levels.

Additional predictors to assess neurocognitive performance will include age, gender, race, degree of carotid stenosis, side of stenosis, prior history of stroke, prior history of neurosurgical or endovascular interventions, presence of coronary artery disease, active malignancy, vasculopathy including diabetes, hypertension, hyperlipidemia, obesity, systemic vascular disease, intracranial atherosclerosis, ultrasound perfusion of intracranial vessels, prior neurocognitive decline: ie prior history of Alzheimer's, degenerative neurological disease. Outcome variables will include standardized neuropsychological measures. The investigators hypothesize a more exuberant neurocognitive response in patients with an incomplete circle of Willis.

A dropped model will be performed to prevent overfitting of the regression analysis. A p value less than 0.05 will be used to define statistical significance.

The investigators predict that patients will not have a statistically significant change in neurocognitive performance during the three-month and six-week time points prior to intervention-and this will serve as the control period. We predict that 35% of patients will have some improvement in neurocognition after intervention. The sample size calculator to identify a difference in groups at a p<0.05 with a power of 0.8 predicts with 5% attrition determines that 20 patients will be required for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years of age
* ultrasound evidence of carotid stenosis; in which the patient has either 50% or greater symptomatic carotid stenosis or 70% or greater asymptomatic carotid stenosis.

Exclusion Criteria:

1. patients <18 years of age
2. patients with without compatibility for MRI
3. patients requiring carotid stenting for reasons not related to long-standing stenosis
4. patients requiring emergency carotid stenting for acute symptoms such as crescendo transient ischemic attacks, intolerance of physiologic blood pressure.
5. Patients that do not have appropriate capacity (i.e. understand the risks and benefits associated with this study) or are unable to consent for themselves will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neurocognition | 4 months
  Neurocognition will be assessed through a battery of 8 tests to measure cognitive capacity across a range of neurocognitive domains.

SECONDARY OUTCOMES:
TNF-α | 4 months
  Inflammatory Markers: tumor necrosis factor-α
IL-6 | 4 months
  Inflammatory Markers: IL-6
IL-1β | 4 months
  Inflammatory Markers: IL-1β
CRP | 4 months
  Inflammatory Markers: CRP
IFN-γ | 4 months
  Inflammatory Markers: IFN-γ
sICAM-1 | 4 months
  Inflammatory Markers: sICAM-1
sVCAM-1 | 4 months
  Inflammatory Markers: sVCAM-1

CONTACTS AND LOCATIONS:
Overall Officials: Alexander A Khalessi, MD, Principal Investigator — UC San Diego; David R Santiago-Dieppa, MD, Study Director — UC San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Per institutional review board, data will only be shared with the researchers specified on the research protocol.

REFERENCES:
- [Background] Arntzen KA, Schirmer H, Johnsen SH, Wilsgaard T, Mathiesen EB. Carotid atherosclerosis predicts lower cognitive test results: a 7-year follow-up study of 4,371 stroke-free subjects - the Tromso study. Cerebrovasc Dis. 2012;33(2):159-65. doi: 10.1159/000334182. Epub 2012 Jan 5. PMID 22222422
- [Background] Baracchini C, Mazzalai F, Gruppo M, Lorenzetti R, Ermani M, Ballotta E. Carotid endarterectomy protects elderly patients from cognitive decline: a prospective study. Surgery. 2012 Jan;151(1):99-106. doi: 10.1016/j.surg.2011.06.031. Epub 2011 Sep 22. PMID 21943640
- [Background] Shapiro AM, Benedict RH, Schretlen D, Brandt J. Construct and concurrent validity of the Hopkins Verbal Learning Test-revised. Clin Neuropsychol. 1999 Aug;13(3):348-58. doi: 10.1076/clin.13.3.348.1749. PMID 10726605
- [Background] Blake GJ, Ridker PM. Novel clinical markers of vascular wall inflammation. Circ Res. 2001 Oct 26;89(9):763-71. doi: 10.1161/hh2101.099270. PMID 11679405
- [Background] Cheng Y, Wang YJ, Yan JC, Zhou R, Zhou HD. Effects of carotid artery stenting on cognitive function in patients with mild cognitive impairment and carotid stenosis. Exp Ther Med. 2013 Apr;5(4):1019-1024. doi: 10.3892/etm.2013.954. Epub 2013 Feb 8. PMID 23596467
- [Background] North American Symptomatic Carotid Endarterectomy Trial Collaborators; Barnett HJM, Taylor DW, Haynes RB, Sackett DL, Peerless SJ, Ferguson GG, Fox AJ, Rankin RN, Hachinski VC, Wiebers DO, Eliasziw M. Beneficial effect of carotid endarterectomy in symptomatic patients with high-grade carotid stenosis. N Engl J Med. 1991 Aug 15;325(7):445-53. doi: 10.1056/NEJM199108153250701. PMID 1852179
- [Background] Wendell CR, Waldstein SR, Ferrucci L, O'Brien RJ, Strait JB, Zonderman AB. Carotid atherosclerosis and prospective risk of dementia. Stroke. 2012 Dec;43(12):3319-24. doi: 10.1161/STROKEAHA.112.672527. Epub 2012 Oct 25. PMID 23103489
- [Background] Sun Q, Xia Z, Qu C, Ruan X, Li J, Cong L, Zheng X, Du Y. Carotid artery stenting ameliorates the cognitive impairment in patients with leukoaraiosis, the ischemic change of cerebral white matter. Tohoku J Exp Med. 2014 Aug;233(4):257-64. doi: 10.1620/tjem.233.257. PMID 25098321